CLINICAL TRIAL: NCT01934699
Title: Intraprocedural Determination of Myocardial Vitality Using Speckle Tracking Echocardiography Compared to Two-time MRI Diagnostics
Brief Title: Intraprocedural Determination of Myocardial Vitality Using 2 Different Imaging Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-004; 00012377 (Other: DIMDI-Nr.)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Angina Pectoris; Left Ventricular Wall Motion Abnormalities
Keywords: Coronary stenosis; Angina pectoris; Left ventricular wall motion abnormalities; 2D-Strain
MeSH Terms: conditions — Angina Pectoris; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI-Arm (Active Comparator): Myocardial vitality determination based on MRI diagnostics.
  Interventions: Device: MRI scanner
- Echo-Arm (Experimental): Myocardial vitality determination using echocardiography in combination with 2D-Strain Analysis.
  Interventions: Device: Cardiac ultrasound

INTERVENTIONS:
Device: Cardiac ultrasound — Patient will get echocardiographic examination during coronary angiography. 2D-Strain Analysis will be performed based on data of these echocardiographic examination. Only when vitality in the contraction impaired segments will be established based on 2D-Strain Analysis, PCI will be performed.
  Arms: Echo-Arm
Device: MRI scanner — Coronary angiography on patient will be canceled. Patients will get viability assessment using MRI within the next 7 days. When vitality will be established with MRI, patient will get PCI.
  Arms: MRI-Arm

SUMMARY:
The investigators will compare myocard vitality diagnostics using 2D-Strain echography and MRI.

DETAILED DESCRIPTION:
Each patient with typical angina pectoris symptoms will get echocardiographic examination during the inclusion phase. If motion disorder of regional left ventricular myocardial wall is detected, patient will get coronary angiography (not study related, caused of typical angina pectoris symptoms and high probability of CHD). If coronary stenosis related to motion disorder is available, patient will be randomized in two groups during coronary angiography.

* First Group: Patient will get echocardiographic examination during coronary angiography. 2D-Strain Analysis will be performed based on data of this echocardiographic examination. Only when vitality in the contraction impaired segments will be established based on 2D-Strain Analysis, PCI (Percutaneous Coronary Intervention) will be performed.
* Second Group: Coronary angiography by patient will be canceled. Patients will get viability assessment using MRI(Magnetic resonance imaging) within the next 7 days. When vitality will be established with MRI, patient will get PCI (Percutaneous Coronary Intervention).

In addition, as part of a feasibility analysis, the possibility of a consolidation of data of coronary angiography with the ultrasound images will be researched by first group of patients. The aim is to simplify the visualization of the intraprocedural vitality detection. For this purpose, a position sensor based on electromagnetic fields (EMT) will be used during coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Typical angina pectoris symptoms
* Echocardiographic determination of regional motion disfunction of left ventricular wall
* Establishment of needly treatment of stenosis related to motion disorder based on coronar angiography.
* Feasibility of MRI-Examination.
* Patients which are legally competent and which are mentally able to understand the study staff
* Patients give their written consent

Exclusion Criteria:

* Allergy against contrast agent
* Patients with limited renal function(GFR < 60 ml/min)
* Acute or instable angina pectoris

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
State of health score | 6 month after diagnistics
  State of health score will be determinated by all patients for the evaluation of clinical outcomes (using the standardized questionnaire on state of health (SF-36))6 months after clinical diagnostics.

SECONDARY OUTCOMES:
Left ventricular function (ejection function) | 6 month after diagnistics
  Left ventricular function (ejection function) by all patients will be determinated 6 month after diagnostics.
End-diastolic and end-systolic volume. | 6 month after diagnostics
  End-diastolic and end-systolic volume will be determined by all patients 6 month after diagnostics
Capture of Major Adverse Cardiac and Cerebrovascular Events(MACCE) | 18 month after diagnostics
  It will be determined, whether all patients suffered any major adverse cardiac and cerebrovascular events (MACCE) inter alia stroke, myocardial infarction, death 18 month after diagnostics

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, MD, Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany